CLINICAL TRIAL: NCT03198637
Title: Comparison of Neuromuscular Blockade's Monitoring and Clinical Assessment During Cisatracurium Paralysis in Critically Ill Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MONITOR
Record Dates: First submitted 2016-06-10; First posted 2017-06-26 (Actual); Last update posted 2018-05-31 (Actual); Status verified 2018-05

CONDITIONS: Critical Illness
Keywords: efficient; neuromuscular; blockade
MeSH Terms: conditions — Critical Illness

ARMS (2):
- Monitoring (Experimental): Neuromuscular Blockade's monitoring
  Interventions: Drug: Cisatracurium's monitoring by TOF (train-of-four) WATCH device.
- Clinical assessment (Active Comparator): No active monitoring of cisatracurium
  Interventions: Drug: clinical assessment

INTERVENTIONS:
Drug: Cisatracurium's monitoring by TOF (train-of-four) WATCH device. — Neuromuscular blockade's monitoring by Cisatracurium thanks to TOF (train-of-four) WATCH device.
  Arms: Monitoring
Drug: clinical assessment
  Arms: Clinical assessment

SUMMARY:
The main objectives of the prolonged resuscitation paralysis are usually adaptation to mechanical ventilation, lower insufflation pressures and cough suppression.

The use of monitoring during the prolonged neuromuscular blockade is the subject of recommendations. Its interest is subject to a recommendation grade B and its use in prevention of overdose is associated with a recommendation of Grade C.

However, many practitioners continue to objectify the depth of neuromuscular blockade and reversal by simple clinical evaluation. This is a subjective estimate of the depth of neuromuscular block.

Resuscitation in several pharmacokinetic parameters are taken into account. First, the drug distribution volume is usually increased in the Intensive Care patient and requires an increase in initial doses to obtain the same pharmacological effect.

Then, unlike a short-term administration, the administration of neuromuscular blocking agents on days causes diffusion in peripheral compartments. Their diffusion coefficients are slower which contributes to the increase of the elimination period after interruption of the administration of curare. There is therefore a risk of residual paralysis.

Secondarily, the curare needs can be influenced by thermoregulation, water and electrolyte disorders and acid-base, administration of certain drugs, the inter- and intra-individual variability and tachyphylaxis (form tolerance of particularly rapid installation during a few close administration, linked to the proliferation of cholinergic receptors).

The value of monitoring neuromuscular blockade in intensive care is the prevention of overdose and in finding the lowest effective dose.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* Mechanically ventilated patients
* Indication for prescribing curare extended less than 1 day
* Sedation
* Information form waived by family members or surrogates

Exclusion Criteria:

* Pregnancy,
* Curare infusion ongoing
* Neuromuscular disorders
* Dermal alteration
* Allergy to cisatracurium, atracurium, benzene sulfonic acid
* Expected survival of less than 2 days
* Personal or family history of malignant hyperthermia
* No social security
* Patient under enhanced protection
* Patient participating to an other intervention research or participated within 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-04; Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Reduction of individual cumulative dose in mg cisatracurium | through study completion : from 1 to 20 days

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Poitiers, Poitiers, France